CLINICAL TRIAL: NCT03840590
Title: Adenoma Detection Rate Using Artificial Intelligence System in China
Brief Title: Adenoma Detection Rate Using AI System in China
Acronym: SinoAIADR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other); Shanghai Zhongshan Hospital (Other); Tianjin People's Hospital (Other); Tianjin Nankai Hospital (Other)
Responsible Party: Principal Investigator, En-Da Yu, Director of Department of Colorectal Surgery and Vice Director of GI Endoscopy, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SINOCOLO2019B
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Colorectal Neoplasms; Colonic Polyp; Adenoma
Keywords: adenoma detection rate
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps; Adenoma

STUDY DESIGN:
Intervention Model Description: CSK endoscopic diagnosis and treatment system a new system of artificial intelligence. It is manufactured by Tianjin Yujin Limited in China. It is equipped with the endoscopic mainframe and has the access to the endoscopic video and image. When lesion-like objects appear in the real-time video, the system will alarm the examiners by sound.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-assisted Colonoscopy (Experimental): Participants in this arm undergo AI-assisted colonoscopy using CSK AI system.
  Interventions: Device: CSK AI system
- Standard Colonoscopy (Active Comparator): Participants in this arm undergo standard colonoscopy.
  Interventions: Device: Standard Colonoscopy

INTERVENTIONS:
Device: CSK AI system — CSK system is equipped with the endoscopic mainframe and alarms the examiners when suspect lesions appear.
  Arms: AI-assisted Colonoscopy
Device: Standard Colonoscopy — This is the routine examination in nowadays clinical practice. Both the equipment and the procedure are as usual as clinical routine.
  Arms: Standard Colonoscopy

SUMMARY:
The primary aim of this study is

- to explore the usefulness of Artificial Intelligence system in colonoscopy on adenoma detection rate (ADR). Other aims include to explore the data below when Artificial Intelligence is used.

Mean adenomas detected per procedure, MAP Proximal Adenoma detection rate, pADR Polyp detection rate, PDR Proximal polyp detection rate, pPDR Mean polyps detected per procedure, MPP Withdrawal time, WT Cecal intubation rate, CIR Cecal intubation time, CIT

DETAILED DESCRIPTION:
Colorectal cancer is common in China. Most colorectal cancers happen when an adenoma becomes cancerous. Doctors use colonoscopy to look inside the colon and rectum and find adenomas and remove them. Removing adenomas is known to reduce the chances of a person developing colorectal cancers. The ability of colonoscopists finding adenomas varies, and there is a lot of researches into how to improve "adenoma detection rates".

A new AI system, called the CSK endoscopic diagnosis and treatment system has been designed to improve the rate of polyp detection at colonoscopy. Previous tests have shown that there is a significant improvement in detection of adenomas when the system is used. This study will randomize patients coming for colonoscopy to have their procedure performed as usual or as an AI-assisted colonoscopy. The investigators will record polyp and adenoma detection rates, duration of procedure, participant comfort levels, and complications. All patients referred for colonoscopy will be invited in 4 centers, recruiting a total of 800 participants.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for screening, surveillance, or diagnostic colonoscopy
* All patients must be able to give informed consent

Exclusion Criteria:

* Patients with any absolute contraindications to colonoscopy
* Patients with established or suspicion of large bowel obstruction or pseudo-obstruction
* Patients with known colon cancer or polyposis syndromes
* Patients with known colonic strictures
* Patients with known severe diverticular segments (that is likely to impede colonoscope passage)
* Patients with active colitis (ulcerative colitis, Crohn's colitis, diverticulitis, infective colitis)
* Patients lacking capacity to give informed consent
* Pregnancy
* Patients who are on clopidogrel, warfarin, or other new generation anticoagulants who have not stopped this for the procedure.
* Patients who are attending for a therapeutic procedure or assessment of a known lesion

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate, ADR | At the end of the procedure, up to 1 hour.
  ADR refer to the rate of adenoma detection, calculated as the proportion of subjects with at least one adenoma.

SECONDARY OUTCOMES:
Polyp detection rate, PDR | At the end of the procedure, up to 1 hour.
  PDR refer to the rate of polyp detection, calculated as the proportion of subjects with at least one polyp.

CONTACTS AND LOCATIONS:
Overall Officials: En-Da YU, MD, Principal Investigator — Changhai Hospital
Locations (4):
- China (4):
  - Sixth affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Tianjin Nankai Hospital, Tianjin, Tianjin Municipality
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No